CLINICAL TRIAL: NCT04894682
Title: Safety and Long-term Effects of COVID-19 Vaccines in Patients With Lung Cancer or Indeterminate Pulmonary Nodule--A Real World Study
Brief Title: Safety and Long-term Effects of COVID-19 Vaccines in Patients With Pulmonary Tumor
Acronym: CoVac-Lung
Status: Withdrawn | Type: Observational
Why Stopped: Changes of the anti-epidemic policy
Sponsor: Guangdong Provincial People's Hospital (Other)
Responsible Party: Principal Investigator, GuiBin Qiao, Administrative Director, Department of Thoracic Surgery, Guangdong Provincial People's Hospital
Other Study IDs: KY-Q-2021-087-01
Record Dates: First submitted 2021-05-06; First posted 2021-05-20 (Actual); Last update posted 2023-03-17 (Actual); Status verified 2023-03

CONDITIONS: Lung Cancer; Pulmonary Nodule, Solitary; Pulmonary Nodule, Multiple; COVID-19 Pneumonia; Vaccine Adverse Reaction; SARS-CoV-2 Acute Respiratory Disease
MeSH Terms: conditions — Lung Neoplasms; Solitary Pulmonary Nodule; Multiple Pulmonary Nodules

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Vaccinated Case: Pulmonary nodules/lung cancer patients who have been vaccinated against the SARS-CoV-2 (with any type/brand of vaccine)
  Interventions: Biological: Vaccine inoculation against SARS-CoV-2
- Vaccinated Healthy Control: Healthy people who have been vaccinated against the SARS-CoV-2 (with any type/brand of vaccine)
  Interventions: Biological: Vaccine inoculation against SARS-CoV-2
- Unvaccinated Case: Pulmonary nodules/lung cancer patients who are not vaccinated against the SARS-CoV-2

INTERVENTIONS:
Biological: Vaccine inoculation against SARS-CoV-2 — Inoculation with any type of approved vaccines according to the standard or recommended dose
  Groups: Vaccinated Case; Vaccinated Healthy Control

SUMMARY:
The objective of this study is to assess the inoculation-related symptoms and long-term effects of COVID-19 vaccines in patients with lung cancer or pulmonary nodules in a real-world setting. The investigators aim to provide high-quality evidence for the COVID-19 vaccines in cancer/pre-cancer patients, and to address their concern about the safety profile of the newly developed vaccines.

DETAILED DESCRIPTION:
This study will enroll lung cancer/pulmonary nodule patients or healthy people who had undergone standard vaccination procedures against SARS-CoV-2/COVID-19. This observatory study will apply an electronic questionnaire to collect general information and post-vaccination symptoms or adverse events of vaccinated pulmonary nodules/lung cancer patients and healthy control. The researchers will further analyze whether the vaccine will promote the progression of primary tumors/pulmonary nodules through long-term follow-up. The investigators aim to assess the adverse events and long-term impact of COVID-19 vaccines in patients with lung cancer or pulmonary nodules in a real-world setting, to provide high-quality evidence for the COVID-19 vaccines in cancer/pre-cancer patients, and to address their concern about the safety profile of the newly developed vaccines.

ELIGIBILITY:
Inclusion Criteria:

1. Pulmonary nodule/lung cancer patients confirmed by CT or pathological examination, who have been vaccinated against the SARS-CoV-2
2. Pulmonary nodule/lung cancer patients confirmed by CT or pathological examination, who are not vaccinated against the SARS-CoV-2
3. Healthy people who have been vaccinated against the SARS-CoV-2

Exclusion Criteria:

1. Multiple malignancy in other parts of body;
2. Infected with SARS-CoV-2 virus currently or in the past;
3. Refuse to participate in this study.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All participants in the vaccinated case and unvaccinated case group are/were diagnosed with pulmonary nodules by CT scan or lung cancer by pathological examination, and are enrolled by invitation from the patient registry database(established and maintained by Department of Thoracic Surgery, Guangdong Provincial People's Hospital). All participants in the healthy control group are free of any malignant diseases, including indeterminate tumors in any body part, and are enrolled by randomly invitation from the public.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2021-05-04 (Actual); Primary Completion 2021-08-31 (Estimated); Study Completion 2022-05-31 (Estimated)

PRIMARY OUTCOMES:
Occurence rate of vaccination-related adverse effects | Vaccination-related adverse effects are monitored from the time of inoculation, up to 1 month after each inoculation
  Occurence rate of vaccination-related adverse effects in case group and healthy control group
Time to progression of pulmonary nodules | The date of vaccine inoculation to the date of reported progression of pulmonary nodules by CT scan, up to 12 months
  Time calculated from the date of vaccine inoculation to the date of reported progression of pulmonary nodules by CT scan
Time to recurrence of lung cancer | The date of vaccine inoculation to the date of reported recurrence of lung cancer by pathological examination, up to 12 months
  Time calculated from the date of vaccine inoculation to the date of reported recurrence of lung cancer confirmed by pathological examination

SECONDARY OUTCOMES:
Duration of vaccination-related adverse effects | Vaccination-related adverse events are monitored from the time of inoculation, up to 1 month after each inoculation
  The period of time calculated from the occurrence of vaccination-related adverse effects to the time of remission
Severity of vaccination-related adverse effects | Vaccination-related adverse events are monitored from the time of inoculation, up to 1 month after each inoculation
  The severity of vaccination-related adverse effects is defined as three grades: Grade 1 (self-remission without any intervention); Grade 2 (Remission only after medical intervention/s); Grade 3 (Adverse event-related Hospitalization)

CONTACTS AND LOCATIONS:
Locations (1):
- Guangdong Provincial People's Hospital, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes
Raw anonymized data are available from corresponding investigator upon reasonable request.
Supporting Information: Study Protocol, SAP
Time Frame: Immediately after the completion of study/publication of results, and will be available for 2 years.
Access Criteria: For pooled study or meta-analysis only.